CLINICAL TRIAL: NCT05179512
Title: Replication of the INSPIRE Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-INSPIRE
Record Dates: First submitted 2021-09-20; First posted 2022-01-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tiotropium: Reference group
  Interventions: Drug: Tiotropium
- Salmeterol/Fluticasone: Exposure group
  Interventions: Drug: salmeterol-fluticasone

INTERVENTIONS:
Drug: Tiotropium — Tiotropium dispensing claim is used as the reference group.
  Groups: Tiotropium
Drug: salmeterol-fluticasone — Salmeterol/Fluticasone dispensing claim is used as the exposure group.
  Groups: Salmeterol/Fluticasone

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-80 years [0,0] days
* Diagnosis of COPD [all available data, 0] days
* Clinical history of at least 1 COPD exacerbation [all available data, -43] days

Exclusion Criteria:

* COPD exacerbation [-42, 0] days
* Asthma, eczema, atopic dermatitis, allergic rhinitis [-180, 0] days
* Known respiratory disorder other than COPD e.g. pulmonary fibrosis or interstitial lung disease (ILD), sarcoidosis, lymphangioleiomyomatosis, primary/pulmonary tuberculosis, cystic fibrosis, pulmonary hypertension/other pulmonary heart disease, lung/pulmonary malignancies, alpha-1 antitrypsin deficiency, pneumoconioses and other lung diseases due to external agents [all available data, 0] days
* Narrow angle glaucoma or prostatic hyperplasia or obstruction of the neck of the bladder [-180, 0] days
* At least one 30-day supply prescription claims for oral alfuzosin, doxazosin, tamsulosin, silodosin, finasteride 5 mg, dutasteride [-180,0] days
* Lung transplant or lung volume reduction surgery (LVRS) [all available data, 0] days
* Daily long term oxygen therapy (LTOT) [all available data, 0] days
* Beta-blockers (except eye drops) [-180, 0] days
* Evidence of alcohol, drug or solvent abuse [-180, 0] days
* Use of salmeterol, tiotropium and fluticasone containing inhaler use [-180, 0] days

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score matched retrospective cohort study design comparing tiotropium to salmeterol. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of SFC or tiotropium inhalers (cohort entry date).
Sampling Method: Non-Probability Sample
Enrollment: 98278 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization exacerbation rate per year | Through study completion or censoring, up to 193 days
  Claims-based algorithm: healthcare utilization exacerbation rate per year

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT05179512/Prot_SAP_000.pdf